CLINICAL TRIAL: NCT05327257
Title: A Feasibility and Pilot Randomized Controlled Double-blind Trial of Intermittent Theta Burst Stimulation (iTBS) Repetitive Transcranial Magnetic Stimulation (rTMS) to Improve Memory in Mild Cognitive Impairment (MCI)
Brief Title: iTBS rTMS in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria I. Lapid, M.D. (Other)
Responsible Party: Sponsor-Investigator, Maria I. Lapid, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 21-010661
Record Dates: First submitted 2022-03-20; First posted 2022-04-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assessor blinded to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- iTBS rTMS Left Dorsolateral Prefrontal Cortex (DLPFC) then Vertex (Experimental): Subjects will receive 10 consecutive days of daily single session of iTBS rTMS for 3.5 minutes per day over the DLPFC in the first treatment period, complete a washout period of 4 weeks then receive 1 session of iTBS rTMS for 3.5 minutes daily over the vertex for 10 consecutive days.
  Interventions: Device: iTBS rTMS
- iTBS rTMS Lateral Parietal Cortex (LPC) then Vertex (Experimental): Subjects will receive 10 consecutive days of daily single session of iTBS rTMS for 3.5 minutes per day over the LPC in the first treatment period, complete a washout period of 4 weeks then receive 1 session of iTBS rTMS for 3.5 minutes daily over the vertex for 10 consecutive days.
  Interventions: Device: iTBS rTMS
- iTBS rTMS Vertex then Left Dorsolateral Prefrontal Cortex (DLPFC) (Experimental): Subjects will receive 1 session of iTBS rTMS for 3.5 minutes daily over the vertex for 10 consecutive days in the first treatment period, complete a washout period of 4 weeks then receive 10 consecutive days of daily single session of iTBS rTMS for 3.5 minutes per day over the DLPFC.
  Interventions: Device: iTBS rTMS
- iTBS rTMS Vertex then Lateral Parietal Cortex (LPC) (Experimental): Subjects will receive 1 session of iTBS rTMS for 3.5 minutes daily over the vertex for 10 consecutive days in the first treatment period, complete a washout period of 4 weeks then receive 10 consecutive days of daily single session of iTBS rTMS for 3.5 minutes per day over the LPC.
  Interventions: Device: iTBS rTMS
- iTBS rTMS Vertex only (Sham Comparator): Cognitively normal and healthy controls will receive 1 session of iTBS rTMS for 3.5 minutes daily over the vertex for 10 consecutive days. The vertex serves as a control as there are no functional improvements in cognition with stimulation of the vertex region.
  Interventions: Device: iTBS rTMS

INTERVENTIONS:
Device: iTBS rTMS — Repetitive transcranial magnetic stimulation (rTMS) intermittent Theta Burst Stimulation (iTBS)

SUMMARY:
The purposes of this research are to test whether it is feasible to administer a treatment protocol called intermittent theta burst stimulation (iTBS) repetitive transcranial magnetic stimulation (rTMS) in adults with mild cognitive impairment (MCI), and to test whether iTBS rTMS treatments can improve memory in mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
To test the feasibility of conducting a 10-day Intermittent Theta Burst Stimulation (iTBS) repetitive Transcranial Magnetic Stimulation (rTMS) protocol twice using a cross-over design in individuals with Mild Cognitive Impairment (MCI), pilot test the study protocol to assess study design, and collect pilot data on the effect of stimulations over 3 different brain regions (left dorsolateral prefrontal cortex (DLPFC), lateral parietal cortex (LPC), vertex) on working memory, new-learning and executive function in MCI. Neuropsychological and sleep measures, functional brain magnetic resonance imaging (fMRI), high density EEG and questionnaires will be performed at 5 timepoints - baseline, post-treatment after first period of 10 daily iTBS rTMS sessions, post-washout period of 4 weeks, post-treatment after cross-over to second period of 10 daily iTBS rTMS sessions, and 4 weeks follow-up post-treatment.

ELIGIBILITY:
Inclusion Criteria

* Must speak English fluently
* Diagnosis of MCI as defined by:

  * Clinical diagnosis by a neurologist
  * Neuropsychological testing support of MCI
  * Meet criteria for MCI
  * Subjective cognitive decline reported by participant and/or an informant
  * Objective memory impairment in one or more cognitive domains for age
  * Essentially preserved general cognitive function
  * Largely intact functional activities
  * Does not meet criteria for dementia as judged by a clinician
* Eligible for transcranial magnetic stimulation (TMS) based on safety criteria
* Clinical Dementia Rating=0.5
* Geriatric Depression Scale score less than 6
* Medically stable and in good general health
* Not pregnant, lactating, or of childbearing potential
* Stable medication regimen for at least 4 weeks prior to baseline visit
* Adequate visual and auditory abilities to complete neuropsychological testing
* Ability to provide informed consent
* Have a care partner who is available to accompany the participant to study visits for the duration of the protocol.

Exclusion Criteria

* Inability to communicate in the English language
* Meet criteria for dementia
* Contraindications to TMS or MRI, including patients who have

  * conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or within 30 cm of the treatment coil (e.g., cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments or jewelry)
  * active or inactive implants, including deep brain stimulators, cochlear implants, vagus nerve stimulators or implanted device leads
* Any true positive findings on the TMS safety screening form
* Prior exposure to TMS, electroconvulsive therapy (ECT), or any neurostimulation within the past 12 months
* History of epilepsy or seizures
* Medical conditions that increase risk of seizures

  * History of traumatic brain injury
  * History of intracranial mass or lesion
  * History of stroke, including hemorrhagic stroke and ischemic stroke
* Psychiatric disorders

  * Primary psychotic disorder (schizophrenia, schizoaffective, or schizophreniform disorder), any history
  * Primary mood disorder (major depressive disorder, bipolar disorder) within the past 12 months
  * Substance use disorder (except caffeine and nicotine) within the past 12 months
* Active symptoms of depression, anxiety, mania, psychosis, or substance use (except caffeine and nicotine) within the past year

  * Active symptoms of depression will be identified based on geriatric depression scale ≥ 6
  * Other active symptoms of psychiatric conditions to be determined by study investigators
* Sleep disorders that are considered clinically significant and not sufficiently treated by the investigative team, including untreated obstructive sleep apnea (apnea-hypopnea index >15), untreated/suboptimally treated REM sleep behavior disorder, untreated/suboptimally treated restless legs syndrome
* Pregnancy or suspected pregnancy
* Participation in another concurrent interventional clinical trial
* Any unstable medical condition
* Inability to provide informed consent
* Inability to adhere to the protocol

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Clinician Referrals | 16 weeks
  Total number of participants referred to the study by clinicians
Participant enrollment | 16 weeks
  Total number of participants enrolled in the study
Treatment adherence | 16 weeks
  Total number of participants to comply with all study procedures as identified in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Lapid, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lapid MI, Pagali SR, Basso MR, Croarkin PE, Geske JR, Huston J 3rd, Islam K, Joseph B, Kennebeck WW, Kang D, Kung S, LeMahieu AM, Lundstrom BN, Petersen RC, Sarran MM, Shu Y, Swanson IM, Louis EKS, Wang MK, Varatharajah Y, Wagh N, Welker KM, Worrell GA, Boeve BF. A pilot randomized controlled double-blind trial of intermittent theta burst stimulation (iTBS) repetitive transcranial magnetic stimulation (rTMS) to improve memory in mild cognitive impairment (MCI): a study protocol. Pilot Feasibility Stud. 2025 Apr 1;11(1):35. doi: 10.1186/s40814-025-01625-5. PMID 40170189
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials